CLINICAL TRIAL: NCT03602755
Title: Retrospective Study of the First-line Treatment of Patients With Newly Diagnosed Transplant-ineligible Multiple Myeloma Between 2012 and 2016, Treated According to Routine Clinical Practice in Spain
Brief Title: A Study of the First-line Treatment of Patients With Newly Diagnosed Transplant-ineligible Multiple Myeloma in Spain
Acronym: RETRO
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NDS-MM-002; U1111-1215-4398 (Other: WHO)
Record Dates: First submitted 2018-06-26; First posted 2018-07-27 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: Transplant; Multiple Myeloma; Spain
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with newly diagnosed transplant-ineligible MM: Adult Patients with newly diagnosed MM who were not suitable candidates for ASCT who started first-line treatment for the study disease in a routine clinical practice setting between 2012 and 2016, inclusive.

SUMMARY:
This is an observational, post-authorization, retrospective, multicenter study (PAS-OD) that will be conducted in approximately 20 centers in Spain. In all cases, only data recorded prior to the date of study start will be collected to ensure its retrospective nature, thus reflecting real clinical practice, avoiding any influence on the physician's clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with newly diagnosed MM who were not suitable candidates for ASCT who started anti-myeloma treatment between 2012 and 2016, inclusive.
* Patients who give informed consent before data collection begins.

Exclusion Criteria:

* Patients who participated in a clinical trial for first-line treatment of MM during the study period.
* Patients who are alive, but do not give their IC.
* Patients with MM who did not receive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total, 400 patients with a de novo diagnosis of multiple myeloma who were not suitable candidates for ASCT who started anti-myeloma treatment between 2012 and 2016, inclusive, in a routine clinical practice setting in Spain, will be included.
Sampling Method: Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Description of the first-line treatment regimens | Up to approximately 5 months
  Number of patients in the different first-line treatment regimens, in terms of the main drug used in patients diagnosed de novo with MM who were not candidates for autologous stem cell transplantation (ASCT)

SECONDARY OUTCOMES:
Description of the characteristics of patients with a diagnosis of MM who were not candidates for ASCT in Spain | Up to approximately 5 months
  Number of patients with a diagnosis of MM who were not candidates for ASCT in Spain in each staging group: Stage I, II and III (ISS) and ISS R
Description of the characteristics of patients with a diagnosis of MM who were not candidates for ASCT in Spain | Up to approximately 5 months
  Number of patients with a diagnosis of MM who were not candidates for ASCT in Spain in each MM subtype group
Progression-free survival (PFS) | Up to approximately 5 months
  Is described as time from start of treatment until disease progression or death
Overall survival (OS) | Up to approximately 5 months
  Is described as time from start of the treatment until death
Overall response rate | Up to approximately 5 months
  Is based on IMWG criteria
Duration of response | Up to approximately 5 months
  Is described as time from start of the treatment until end of first line treatment
Patients who receive second-line treatment | Up to approximately 5 months
  Proportion of patients who receive second-line treatment
Patients who underwent dose adjustment or switched treatment | Up to approximately 5 months
  Proportion of patients who underwent dose adjustment or switched treatment
Patients who discontinued treatment | Up to approximately 5 months
  Proportion of patients who discontinued treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Lostaunau, MD, Study Director — Celgene
Locations (20):
- Spain (20):
  - H. Santiago (CHUS), Santiago de Compostela, A Coruña
  - H. Txagorritxu, Vitoria-Gasteiz, Alava
  - H. Son Espases, Palma, Balearic Islands
  - ICO Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - H. Althaia, Manresa, Barcelona
  - H. Mutua de Terrassa, Terrassa, Barcelona
  - H. Jerez, Jerez de la Frontera, Cadiz
  - H. Alvaro Cunqueiro, Vigo, Pontevedra
  - H. Cabueñes, Gijón, Principality of Asturias
  - H. Central de Asturias, Oviedo, Principality of Asturias
  - H. del Mar, Barcelona
  - H. Josep Trueta, Girona
  - H. Arnau de Villanova, Lleida
  - H- Virgen de la Victoria, Málaga
  - H. Carlos Haya, Málaga
  - H. Ourense (CHOU), Ourense
  - H. Virgen Macarena, Seville
  - H. Joan XXIII, Tarragona
  - H. Dr. Peset, Valencia
  - H. La Fe, Valencia